CLINICAL TRIAL: NCT02190006
Title: Comparison Between the Role of Follicular Output Rate and Preovulatory Count in the Prediction of Pregnancy in Women With Polycystic Ovarian Syndrome Undergoing Intra Cytoplasmic Sperm Injection (ICSI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer, Cairo University
Other Study IDs: sub 4
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Polycystic Ovarian Syndrome; Subfertility; ICSI
Keywords: Polycystic ovarian syndrome; Follicle output rate; preovulatory count; ICSI
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Polycystic ovarian syndrome: Women with polycystic ovarian syndrome undergoing ICSI

SUMMARY:
Our study is observational, we are observing data from routine measurements during IVF/ICSI. Our study does not assess IVF/ICSI as an intervention, we are evaluating the role of FSI and preovulatory count which are calculated by observing routine measurements during the IVF/ICSI procedure.

300 women with polycystic ovarian syndrome (PCOS) who are decided to be treated with ICSI. will be subjected to full history taking and clinical examination. On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have standard pituitary down-regulation followed by follicle stimulating hormone (FSH) stimulation until the day of Human chorionic gonadotrophin (HCG) administration.

On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe and the Preovulatory follicle count (PC) will be assessed, (PFC) is defined as number of follicles measuring≥16mm. Follicular output rate (FORT) will be calculated as: (FSI =PFC*10000/AFC*Total dose of FSH).

FORT correlation to pregnancy will be compared to that of the preovulatory count number

DETAILED DESCRIPTION:
Our study is observational, we are observing data from routine measurements during IVF/ICSI. Our study does not assess IVF/ICSI as an intervention, we are evaluating the role of FSI and preovulatory count which are calculated by observing routine measurements during the IVF/ICSI procedure.

All women fulfilling the inclusion criteria will be invited to participate in the study. A written informed consent will be taken and only women signing the consent will be included in the study. Patients included in the study will be subjected to full history taking and clinical examination including general, abdominal and gynecological examination. This will be followed by a vaginal ultrasound scan to assess uterus, ovaries and any pelvic masses.

All women will go through the usual IVF/ICSI procedure explained below, our aim is to observe the antral follicle count, the pre-ovulatory count, and calculate the FORT.

On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have standard pituitary down-regulation protocol with GnRHa (Triptorelin 0.1mg, Decapeptyl® Ferring, Germany) day 7 after ovulation of previous cycle or on day 21 of the oral contraceptive cycles. GnRHa will be continued for 2 weeks. FSH (Fostimon ®IBSA) 150-300 IU/day will be administered until the day of HCG administration.

On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe and the Preovulatory follicle count (PC) will be assessed, (PFC) is defined as number of follicles measuring≥16mm. FORT will be calculated as: (PFC) * 100/AFC.

The procedure will be cancelled if less than 3 follicles 16-20 mm in size are present 12 days after starting FSH despite doses reaching 450 IU. The cycle will be also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG. Oocytes will be fertilized either via IVF or ICSI based on the couple's history. Fertilization will be assessed 16-18 h after IVF or ICSI. Embryo transfers will be performed 3 days after oocyte retrieval. No more than three embryos per patient will be transferred; vaginal tablets containing progesterone (Prontogest® IBSA) administered 400 mg/day as luteal support from the day of the oocyte retrieval. Pregnancy will be defined as the appearance of an intrauterine gestational sac by vaginal ultrasound 5 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosed using the Rotterdam criteria
* Age 20-40 years
* Both ovaries are present
* Day 2 FSH <10 mIU/L
* Day 2 Estradiol<50 pg/L

Exclusion Criteria:

* Other causes of subfertility
* Abnormalities affecting the uterine cavity
* Uncontrolled diabetes
* Allergy to gonadotrophins
* Cancelled cycles during the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 300 women with Polycystic ovarian syndrome who are already decided to be treated with ICSI will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | 5 weeks after embryo transfer
  FORT values will be classified into 3 categories: low, medium and high. The proportion of women achieving a clinical pregnancy will be compared among the 3 groups. Correlation of FORT with clinical pregnancy will be compared with the correlation of preovulatory count with pregnancy using a regression analysis. Clinical pregnancy will be defined as the presence of an intra-uterine gestational sac detected by ultrasound scanning.

SECONDARY OUTCOMES:
Number of embryos | 3 days after embryo transfer
  Correlation between FORT and the number of embryos will be compared to the correlation of preovulatory count and the number of embryos using regression analysis.
Quality of embryos | 3 days after ovum pick up
  The correlation between FORT and the quality of embryos will be compared with the correlation of preovulatory count and the quality of embryos using regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - Dar AlTeb subfertility centre, Giza

REFERENCES:
- [Background] Kar S. Clomiphene citrate or letrozole as first-line ovulation induction drug in infertile PCOS women: A prospective randomized trial. J Hum Reprod Sci. 2012 Sep;5(3):262-5. doi: 10.4103/0974-1208.106338. PMID 23531705
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Kamath MS, George K. Letrozole or clomiphene citrate as first line for anovulatory infertility: a debate. Reprod Biol Endocrinol. 2011 Jun 21;9:86. doi: 10.1186/1477-7827-9-86. PMID 21693034
- [Background] Zhang N, Hao CF, Zhuang LL, Liu XY, Gu HF, Liu S, Chen ZJ. Prediction of IVF/ICSI outcome based on the follicular output rate. Reprod Biomed Online. 2013 Aug;27(2):147-53. doi: 10.1016/j.rbmo.2013.04.012. Epub 2013 May 4. PMID 23768619
- [Background] de Carvalho BR, Rosa e Silva AC, Rosa e Silva JC, dos Reis RM, Ferriani RA, Silva de Sa MF. Ovarian reserve evaluation: state of the art. J Assist Reprod Genet. 2008 Jul;25(7):311-22. doi: 10.1007/s10815-008-9241-2. Epub 2008 Aug 5. PMID 18679790
- [Background] Broer SL, Mol BW, Hendriks D, Broekmans FJ. The role of antimullerian hormone in prediction of outcome after IVF: comparison with the antral follicle count. Fertil Steril. 2009 Mar;91(3):705-14. doi: 10.1016/j.fertnstert.2007.12.013. Epub 2008 Mar 5. PMID 18321493
- [Background] Melo MA, Garrido N, Alvarez C, Bellver J, Meseguer M, Pellicer A, Remohi J. Antral follicle count (AFC) can be used in the prediction of ovarian response but cannot predict the oocyte/embryo quality or the in vitro fertilization outcome in an egg donation program. Fertil Steril. 2009 Jan;91(1):148-56. doi: 10.1016/j.fertnstert.2007.11.042. Epub 2008 May 2. PMID 18455166
- [Background] Genro VK, Grynberg M, Scheffer JB, Roux I, Frydman R, Fanchin R. Serum anti-Mullerian hormone levels are negatively related to Follicular Output RaTe (FORT) in normo-cycling women undergoing controlled ovarian hyperstimulation. Hum Reprod. 2011 Mar;26(3):671-7. doi: 10.1093/humrep/deq361. Epub 2010 Dec 21. PMID 21177311
- [Background] Gallot V, Berwanger da Silva AL, Genro V, Grynberg M, Frydman N, Fanchin R. Antral follicle responsiveness to follicle-stimulating hormone administration assessed by the Follicular Output RaTe (FORT) may predict in vitro fertilization-embryo transfer outcome. Hum Reprod. 2012 Apr;27(4):1066-72. doi: 10.1093/humrep/der479. Epub 2012 Jan 24. PMID 22279090